CLINICAL TRIAL: NCT00997672
Title: A Double-blind, Randomized, Placebo-controlled Clinical Trial to Assess Efficacy, Safety and Tolerability of Lithium in Multiple System Atrophy.
Brief Title: Lithium in Multiple System Atrophy
Acronym: LAMU
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Data Monitoring Committee decision on 22nd August 2011 for safety issues
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Alessandro Filla, Principal Investigator, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSA_LITIO_13; Eudract n°2009-016377-15
Record Dates: First submitted 2009-10-16; First posted 2009-10-19 (Estimated); Results first posted 2014-02-03 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2013-12

CONDITIONS: Multiple System Atrophy
Keywords: MSA; Lithium; Lithium carbonate; MSA-P; MSA-C
MeSH Terms: conditions — Multiple System Atrophy | interventions — Lithium Carbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lithium CARBONATE 150 and/or 300 mg (Experimental)
  Interventions: Drug: Lithium Carbonate
- Placebo (Placebo Comparator): Placebo comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lithium Carbonate — Lithium Carbonate will be dosed based on lithiemy, which will be in the range 0.9-1.2 mEq/L. Maximum allowed dose will be 1500mg/day.
  Arms: Lithium CARBONATE 150 and/or 300 mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine safety and tolerability of the treatment with lithium in Multiple System Atrophy. Moreover, clinical symptoms, neuronal loss, quality of life and depressive symptoms, will be considered to further investigate the effect of lithium therapy.

DETAILED DESCRIPTION:
Patients will be progressively enrolled in the study and undergo a screening visit to test for inclusion/exclusion criteria. Patients will then be randomized to receive either Lithium carbonate or placebo. Patients will visit study center at 2, 4, 8, 12, 24, 36 and 48 weeks, for endpoint and laboratory assessments.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of probable MSA (Gilman, et al. 2008)
* Age ≥18, <80

Exclusion Criteria:

* Heart failure
* Liver disease
* Kidney failure
* Thyroid disease
* Sick sinus syndrome and/or significant ECG alterations
* Hyposodemia
* Treatment with diuretics
* Treatment with haloperidol and/or other antipsychotics
* Treatment with NSAIDs or corticosteroids
* Treatment with ACE inhibitors
* Treatment with aminophyllines
* Treatment with mannitol
* Pregnancy and/or breastfeeding
* Acute diseases that might interfere with the trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Filla, MD, Principal Investigator — University Federico II
Locations (1):
- Dipartimento di Scienze Neurologiche, Napoli, Italy

REFERENCES:
- [Background] Gilman S, Wenning GK, Low PA, Brooks DJ, Mathias CJ, Trojanowski JQ, Wood NW, Colosimo C, Durr A, Fowler CJ, Kaufmann H, Klockgether T, Lees A, Poewe W, Quinn N, Revesz T, Robertson D, Sandroni P, Seppi K, Vidailhet M. Second consensus statement on the diagnosis of multiple system atrophy. Neurology. 2008 Aug 26;71(9):670-6. doi: 10.1212/01.wnl.0000324625.00404.15. PMID 18725592
- See also: University Federico II — http://www.unina.it
- See also: AOU Policlinico "Federico II" — http://www.policlinico.unina.it

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited through our outpatient clinic. Recruitment started the 4th June 2010 and the trial was stopped the 22nd of August 2011
Pre-assignment Details: Patients were screened prior to randomization, no patients were excluded.
Groups:
- Lithium CARBONATE 150 or 300 mg: Lithium Carbonate : Lithium Carbonate will be dosed based on lithiemy, which will be in the range 0.9-1.2 mEq/L. Maximum allowed dose will be 1500mg/day.
- Placebo: Placebo
Period: Overall Study
Arm/Group | Lithium CARBONATE 150 or 300 mg | Placebo
Started | 4 | 5
Completed | 0 | 1
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Lithium Carbonate : Lithium Carbonate will be dosed based on lithiemy, which will be in the range 0.9-1.2 mEq/L. Maximum allowed dose will be 1500mg/day.
- Total: Total of all reporting groups
Arm/Group | Lithium CARBONATE 150 or 300 mg | Placebo | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 4 | 6
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (5) | 64 (6) | 64 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  Italy | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Primary Endpoint of the Study Will be the Difference in Number and Relative Frequency of Severe Adverse Events (SAE) and Non Severe Adverse Events (nSAE) Recorded During the Study, Between Treatment and Placebo Group.
Description: Number of Adverse Events and their relative frequency in treatment groups was analyzed
Time Frame: the endpoint will be recorded at all visits
Measure: Number; unit: number of AEs
Arm/Group | Lithium CARBONATE 150 or 300 mg | Placebo
Number analyzed (Participants) | 4 | 5
number of AEs | 58 | 21

2. Secondary Outcome: Secondary Outcome Will be the Unified Multiple System Atrophy Rating Scale (UMSARS). Statistical Analysis Will be Performed to Compare the Effect of Treatment on Both Groups.
Time Frame: 0 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Micro- and Macrostructural Magnetic Resonance Parameters Will be Compared Before and After Treatment. This Will Include Voxel Based Morphometry, Resting Functional MRI, Diffusion Tensor Imaging and MRI Spectroscopy.
Time Frame: 0 weeks
Reporting Status: Not Posted

4. Secondary Outcome: The Effect of Lithium on Mood Will be Explored With the Beck Depression Inventory.
Time Frame: 0 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Effect of Lithium on Quality of Life Will be Assessed With the EQ-5D Scale.
Time Frame: 0 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Secondary Outcome Will be the Unified Multiple System Atrophy Rating Scale (UMSARS). Statistical Analysis Will be Performed to Compare the Effect of Treatment on Both Groups.
Time Frame: 24 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Secondary Outcome Will be the Unified Multiple System Atrophy Rating Scale (UMSARS). Statistical Analysis Will be Performed to Compare the Effect of Treatment on Both Groups.
Time Frame: 48 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Micro- and Macrostructural Magnetic Resonance Parameters Will be Compared Before and After Treatment. This Will Include Voxel Based Morphometry, Resting Functional MRI, Diffusion Tensor Imaging and MRI Spectroscopy.
Time Frame: 48 weeks
Reporting Status: Not Posted

9. Secondary Outcome: The Effect of Lithium on Mood Will be Explored With the Beck Depression Inventory.
Time Frame: 24 weeks
Reporting Status: Not Posted

10. Secondary Outcome: The Effect of Lithium on Mood Will be Explored With the Beck Depression Inventory.
Time Frame: 48 weeks
Reporting Status: Not Posted

11. Secondary Outcome: Effect of Lithium on Quality of Life Will be Assessed With the EQ-5D Scale.
Time Frame: 24 weeks
Reporting Status: Not Posted

12. Secondary Outcome: Effect of Lithium on Quality of Life Will be Assessed With the EQ-5D Scale.
Time Frame: 48 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Lithium CARBONATE 150 or 300 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 4/4 | 1/5
Other Adverse Events (participants affected / at risk) | 4/4 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lithium CARBONATE 150 or 300 mg (N=4) | Placebo (N=5)
Death (Cardiac disorders) | 1 (1) | 1 (1)
Cardiovascular failure (Cardiac disorders) | 1 (1) | 1 (1)
Pulmonary infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fever (Infections and infestations) | 1 (1) | 0 (0)
Inguinal abscess (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lithium CARBONATE 150 or 300 mg (N=4) | Placebo (N=5)
Lower limbs weakness (Nervous system disorders) | 3 (4) | 3 (5)
sleepiness (Nervous system disorders) | 1 (4) | 2 (5)
Incontinence (Renal and urinary disorders) | 1 (4) | 3 (5)
Cystitis (Renal and urinary disorders) | 2 (4) | 1 (5)
diarrhea (Gastrointestinal disorders) | 2 (4) | 2 (5)
joint rigidity (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (5)
pulmonitis (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 1 (5)
gastroaesophageal reflux (Gastrointestinal disorders) | 1 (4) | 2 (5)

LIMITATIONS AND CAVEATS:
Limitation of the study is small sample size of nine randomized patients. This may have determined uneven distribution of AEs due to random variation. Taking into account these limitations, we do not encourage future studies with lithium in MSA.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No